CLINICAL TRIAL: NCT02501460
Title: Impact of Resistance Training-Protein Supplementation on Lean Muscle Mass in Childhood Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: ATC Fitness (Unknown); American Institute for Cancer Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: REPS; AICR FDN YR 1 (Other Grant/Funding Number: American Institute for Cancer Research); NCI-2015-01152 (Registry Identifier: NCI Clinical Trial Registration Program)
Record Dates: First submitted 2015-07-15; First posted 2015-07-17 (Estimated); Last update posted 2018-07-17 (Actual); Status verified 2018-07

CONDITIONS: Cancer
Keywords: Adult cancer survivors; Exercise; Dietary supplementation
MeSH Terms: conditions — Neoplasms; Motor Activity | interventions — Guidelines as Topic; Resistance Training; Exercise; Dietary Supplements

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supplement Group (Active Comparator): Participants will receive educational handouts and complete research testing to evaluate their physical condition prior to beginning the resistance training and dietary supplementation. Adherence will be assured as described below.
  Interventions: Other: Educational handouts; Other: Resistance training; Dietary Supplement: Supplementation
- Placebo Group (Placebo Comparator): Participants will receive educational handouts and complete research testing to evaluate their physical condition prior to beginning the resistance training and placebo. Adherence will be assured as described below.
  Interventions: Other: Educational handouts; Other: Resistance training; Other: Placebo

INTERVENTIONS:
Other: Educational handouts — Both groups of participants will receive educational handouts that explain the Physical Activity Guidelines for Americans at enrollment.
  Other Names: guidelines
Other: Resistance training — Individuals in both groups will participate in an individually tailored progressive resistance training program 3 times/week for 24 weeks. During weeks 1-4 participants will be supervised twice a week tapering to once a week in weeks 5-12, every other week in weeks 13-20 and then once a month in weeks 21-24 by an American College of Sports Medicine (ACSM) Certified Exercise Specialist (trainer).
  Adherence: To assure fidelity and safety of the resistance training component of the intervention, participants will initially be supervised more frequently They will complete an exercise log for each of their sessions. As the supervision level for exercise is tapered, participants may receive reminders to exercise and take their supplement/placebo via text, phone, or e-mail as needed.
  Other Names: exercise
Dietary Supplement: Supplementation — A medical quality protein supplement powder will be mixed with water or a sugar free drink mix to be taken daily within 60 minutes of training on exercise days or mid-morning on non-exercise days.
  Other Names: protein dietary supplement
  Arms: Supplement Group
Other: Placebo — A placebo that appears to be identical to the medical quality protein supplement powder will be mixed with water or a sugar free drink mix to be taken daily within 60 minutes of training on exercise days or mid-morning on non-exercise days.
  Arms: Placebo Group

SUMMARY:
This study is being conducted because low lean muscle mass is prevalent among childhood cancer survivors. Lean muscle is the non-fatty muscle tissue that makes up part of the body's lean body mass. Low lean muscle mass is associated with loss of overall body strength, declining mobility and eventually, loss of independence. Among childhood cancer survivors, low lean muscle mass may contribute to reduced physical functioning and a sense of fatigue with exertion, limiting ability to participate in adequate physical activity. Loss of strength and a sense of fatigue with repeated movement make it difficult to participate in daily activities.

Although there have not been exercise intervention studies among childhood cancer survivors specifically designed to evaluate the effects of resistance training on muscle mass, studies among individuals with chronic disease, including survivors of adult onset cancers, indicate that resistance exercise improves muscle mass, muscle strength, mobility, vitality and physical activity levels. Resistance training (weight lifting) is a form of physical activity that is designed to improve muscular fitness by exercising a muscle or a muscle group against external resistance.

The purpose of the study is to evaluate the effects of resistance training combined with either a protein supplement or a sports drink on changes in lean muscle mass in young adults who were treated for childhood cancer. The sports drink, for this study, is considered a placebo.

DETAILED DESCRIPTION:
This double-blind placebo controlled study will randomize adult survivors of childhood cancer who are 18 to 44 years of age, greater than ten years post first cancer diagnosis, and with low lean muscle mass to two groups: Resistance Training + Supplement (RT+S) or Resistance Training + Placebo (RT+P). Randomization will be stratified by sex and age (18-29 and 30-44 years) in a block size of 4. Three weekly resistance training sessions will occur over a 24 week period. The participants, investigator, trainer and individuals involved in testing will be blind to group assignment.

Participants will receive information about physical activity and its health benefits. They will be randomly assigned to one of two groups to receive individually tailored resistance training three times per week for 24 weeks. One group will receive a protein supplement, while the other group will receive a sports drink (placebo).

To assess outcomes, participants will have the following research tests:

* Blood will be drawn to assess heart health.
* Questionnaires will be completed to assess physical activity and health as well as food intake.
* Blood pressure measurement.
* Electrocardiogram to assess heart health.
* Height, weight, waist and hip measurements.
* Lean muscle mass will be measured by dual x-ray absorptiometry (DEXA scan).
* Muscle strength will be measured by handgrip, knee extension, and ankle dorsiflexion.
* Walking speed to determine usual walking speed.
* Six-minute walk test to determine endurance.
* Physical activity will be monitored by having the participant complete a survey and wear a small recording device (accelerometer) for seven days.

Study Objectives:

* To evaluate the effects of 24-week supervised RT+S compared to RT+P on changes in lean muscle mass, muscle strength, walking speed, self-reported exhaustion and physical activity levels among childhood cancer survivors.
* To evaluate the effects of 24-week supervised RT+S compared to RT+P on changes in blood pressure, high density lipoprotein, triglycerides, abdominal obesity, fasting glucose, fasting insulin, and C-reactive protein among childhood cancer survivors.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be enrolled on the SJLIFE protocol at St. Jude Children's Research Hospital.
* 18.0-44.99 years of age
* >10 years post first cancer diagnosis.
* English speaking.
* Live within a 45-minute drive of a greater Memphis area ATC Fitness Center
* Low lean mass defined as either:

  * Age- and sex-specific relative lean muscle mass standard deviation score ≤ -1.0.

OR

* Body fat content greater than or equal to 25% in males or greater than or equal to 35% in females.

Exclusion Criteria:

* Currently pregnant (assessed by serum pregnancy test).
* Contraindications to resistance training or protein supplementation (e.g. renal) verified by a physician.

Ages: 18 Years to 44 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 130 (Actual)
Dates: Start 2015-08-17 (Actual); Primary Completion 2018-01-30 (Actual); Study Completion 2018-01-30 (Actual)

PRIMARY OUTCOMES:
Change in lean muscle mass by arm | Baseline and at 24 weeks
  Dual x-ray absorptiometry (DEXA) will be used to determine lean muscle mass. Fat free mass will be measured in the total body scanning mode.
Change in handgrip by arm | Baseline and at 24 weeks
  Handgrip strength will be evaluated with a hand held dynamometer.
Change in knee extension by arm | Baseline and at 24 weeks
  Knee extension strength will be evaluated with the Biodex System IV dynamometer.
Change in ankle dorsiflexion by arm | Baseline and at 24 weeks
  Ankle dorsiflexion strength will be evaluated with the Biodex System IV dynamometer.
Change in walking speed by arm | Baseline and at 24 weeks
  Usual walking speed will be evaluated by having participants complete a timed 10 meter walk test.
Change in endurance by arm | Baseline and at 24 weeks
  Endurance will be evaluated by having participants complete the six minute walk test in a level of corridor as outlined by the American Thoracic Society.
Change in activity level by arm | Baseline and at 24 weeks
  Participants will complete the physical activity monitor (PAM) component of the most recent release of the National Health and Nutrition Examination Survey to measure activity levels. The PAM collects information on intensity and duration of common activities like walking and jogging for seven consecutive days. Participants will receive an accelerometer with written instructions, programmed to begin recording 12:01 a.m. on the day after the baseline assessment (the week before they begin training) and the day after their final training appointment.
Change in blood pressure by arm | Baseline and at 24 weeks
  Blood pressure will be evaluated with a sphygmomanometer.
Change in high density lipoprotein by arm | Baseline and at 24 weeks
  High density lipoprotein will be evaluated from fasting blood samples as part of a standard lipid panel.
Change in triglycerides by arm | Baseline and at 24 weeks
  Triglycerides will be evaluated from fasting blood samples as part of a standard lipid panel.
Change in abdominal obesity by arm | Baseline and at 24 weeks
  Abdominal obesity will be evaluated by measuring waist circumference with a Gulick tape measure to the nearest mm.
Change in fasting glucose by arm | Baseline and at 24 weeks
  Glucose level will be measured from fasting blood samples.
Change in fasting insulin by arm | Baseline and at 24 weeks
  Insulin level will be measure from fasting blood samples.
Change in C-reactive protein by arm | Baseline and at 24 weeks
  Highly sensitive C-reactive protein will be measured from fasting blood samples.
Change in self-reported exhaustion by arm | Baseline and at 24 weeks
  Measured using the vitality subscale of the Medical Outcomes Survey Short Form-36 (SF-36), version 2.

CONTACTS AND LOCATIONS:
Overall Officials: Kirsten K. Ness, PT, PhD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials open at St. Jude — http://www.stjude.org/protocols